CLINICAL TRIAL: NCT04940091
Title: Association Between the Effect of Epidural Analgesia and the Development of Maternal Fever During Labor: a Multicenter, Prospective, Observational, Cohort Study
Brief Title: Epidural Analgesia and Maternal Fever During Labor
Status: Completed | Type: Observational
Sponsor: Peking University First Hospital (Other)
Collaborators: Guangdong Women and Children Hospital (Other); Tangshan Maternal and Child Health Hospital (Other); Dongguan Maternal and Child Health Hospital (Unknown); Beijing Haidian Maternal and Child Health Hospital (Other); Beijing Fuxing Hospital (Unknown); The Fourth Hospital of Shijiazhuang (Other); Xiamen Maternity & Child Care Hospital (Other)
Responsible Party: Principal Investigator, Dong-Xin Wang, Professor, Peking University First Hospital
Other Study IDs: 2021-173
Record Dates: First submitted 2021-06-09; First posted 2021-06-25 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Epidural Analgesia; Analgesic Effect; Fever
Keywords: Epidural labor analgesia; Analgesic effect; Maternal fever during labor
MeSH Terms: conditions — Fever | interventions — Analgesia, Epidural

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 42 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Epidural labor analgesia: All participants will receive epidural analgesia during labor.
  Interventions: Drug: Epidural analgesia

INTERVENTIONS:
Drug: Epidural analgesia — Epidural analgesia is performed with a mixture of local anesthetics (ropivacaine) and opioids (sufentanil).
  Other Names: No other intervention

SUMMARY:
Women who receive epidural analgesia during labor are more likely to develop fever than those who do not. Maternal fever during labor can produce various harmful effects on both mothers and infants. The investigators speculate that the effect of epidural analgesia is associated with the development of maternal fever, i.e., better analgesia is associated with higher risk of maternal fever.

DETAILED DESCRIPTION:
Epidural related maternal fever (ERMF) refers to the phenomenon of increased body temperature of parturient after receiving epidural analgesia during labor. Women who receive epidural labor analgesia are more likely to have fever than those who do not. In a systematic review, 20-33% of parturients receiving neuraxial analgesia developed fever during labor, compared with only 5-7% of those without neuraxial analgesia. Maternal fever can interfere with women's laboring process, decrease the sensitivity of the uterus and cervix to oxytocin, and lead to dystocia and increased surgical delivery rate. The investigators note that the rate of ERMF is lower in patients receiving lower density neuraxial blockade. The study is designed to test the hypothesis that the effect of epidural analgesia is associated with the development of maternal fever, i.e., better analgesia is associated with higher risk of maternal fever.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years old;
* Nulliparae with single term cephalic pregnancy;
* Preparing to give vaginal delivery under epidural analgesia.

Exclusion Criteria:

* Basal body temperature ≥37.3°C;
* Presence of serious pregnancy complications (such as severe preeclampsia, placenta accreta, HELLP [Hemolysis, Elevated Liver enzymes, Low Platelet count] syndrome, placenta previa, abruption of placenta, or hyperthyroidism);
* History of hyperthyrodism, including hyperthyrodism in pregnancy;
* Taking sedatives and/or analgesics within one week before planned delivery;
* American Society of Anesthesiologists classification >class III;
* Contraindications to epidural puncture, including central nervous system diseases (such as poliomyelitis), spinal diseases (such as intraspinal mass, lumbar disc herniation, history of spinal trauma, etc.), abnormal blood coagulation, etc.;
* Presence of infections, including obstetric infections, systemic infections (such as sepsis, bacteremia), or infections at the puncture site or adjacent sites;
* Other conditions that are considered unsuitable for study participation;
* Refused to participate in the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — pregnant women
Study Population: Adult (≥18 years old) nulliparae with single term cephalic pregnancy preparing to give vaginal delivery under epidural analgesia.
Sampling Method: Probability Sample
Enrollment: 1051 (Actual)
Dates: Start 2021-06-10 (Actual); Primary Completion 2022-02-05 (Actual); Study Completion 2022-03-21 (Actual)

PRIMARY OUTCOMES:
Occurrence of maternal fever during labor | delivery ( the end of childbirth.)
  Maternal fever is defined as temperature of ≥38℃ during any stage of labor.

SECONDARY OUTCOMES:
Occurrence of mild maternal fever during labor | delivery ( the end of childbirth.)
  Mild maternal fever is defined as temperature of >37.5℃ during any stage of labor.
Duration of labor | delivery ( the end of childbirth.)
  Duration of the first, second, and third stage of labor.
Neonatal Apgar score | At 1 and 5 minutes after birth.
  Apgar score is assessed at 1 and 5 minutes after birth.
Postpartum hospital stay | Up to 42 days after childbirth.
  Postpartum hospital stay
Postpartum pain intensity | At 1, 10 and 42 days after childbirth
  Pain intensity is assessed with numeric rating scale (NRS; an 11-point scale where 0=no pain and 10=the worst pain).
Postpartum breastfeeding | At 1, 10 and 42 days after childbirth
  The status of breastfeeding include breastfeeding, formula milk, or a mix of them.
Postpartum persistent pain | At 42 days after childbirth
  Defined as NRS pain score ≥1 that persisted since childbirth. For those with persistent pain, also ask if the following activities was affected, including walking, mood, sleep or concentration, as judged by parturients themselves.
Postpartum depression score | At 10 and 42 days postpartum
  Postpartum depression is assessed with the the Edinburgh Postnatal Depression Scale. This is a 10-item self-report questionnaire; each item is rated from 0 to 3 denoting the increasing severity of symptoms, resulting in a maximum score of 30. A score ≥10 is defined as the presence of depression.
Postpartum complications | Up to 42 days postpartum
  Include maternal and neonatal complications, indicate new onset medical events that are harmful and required therapeutic intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Dong-Xin Wang, MD, PhD, Principal Investigator — Peking University First Hospital
Locations (8):
- China (8):
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Xiamen maternal and child hospital, Xiamen, Fujian
  - Dongguan women and children's hospital, Dongguan, Guangdong
  - Guangzhou Women and Children's Medical Center, Guangzhou, Guangdong
  - Shijiazhuang Obstetric and Gynecology Hospital, Shijiazhuang, Hebei
  - Tangshan maternal and child hospital, Tangshan, Hebei
  - Beijing Fuxing Hospital, Beijing
  - Beijing Haidian women and children's Hospital, Beijing

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Arendt KW, Segal BS. The association between epidural labor analgesia and maternal fever. Clin Perinatol. 2013 Sep;40(3):385-98. doi: 10.1016/j.clp.2013.06.002. Epub 2013 Jul 19. PMID 23972746
- [Background] Fusi L, Steer PJ, Maresh MJ, Beard RW. Maternal pyrexia associated with the use of epidural analgesia in labour. Lancet. 1989 Jun 3;1(8649):1250-2. doi: 10.1016/s0140-6736(89)92341-6. PMID 2566791
- [Background] Camann WR, Hortvet LA, Hughes N, Bader AM, Datta S. Maternal temperature regulation during extradural analgesia for labour. Br J Anaesth. 1991 Nov;67(5):565-8. doi: 10.1093/bja/67.5.565. PMID 1751270
- [Background] Lucas MJ, Sharma SK, McIntire DD, Wiley J, Sidawi JE, Ramin SM, Leveno KJ, Cunningham FG. A randomized trial of labor analgesia in women with pregnancy-induced hypertension. Am J Obstet Gynecol. 2001 Oct;185(4):970-5. doi: 10.1067/mob.2001.117970. PMID 11641687
- [Background] Sharma SK, Alexander JM, Messick G, Bloom SL, McIntire DD, Wiley J, Leveno KJ. Cesarean delivery: a randomized trial of epidural analgesia versus intravenous meperidine analgesia during labor in nulliparous women. Anesthesiology. 2002 Mar;96(3):546-51. doi: 10.1097/00000542-200203000-00007. PMID 11873026
- [Background] Sharma SK, Sidawi JE, Ramin SM, Lucas MJ, Leveno KJ, Cunningham FG. Cesarean delivery: a randomized trial of epidural versus patient-controlled meperidine analgesia during labor. Anesthesiology. 1997 Sep;87(3):487-94. doi: 10.1097/00000542-199709000-00006. PMID 9316951
- [Background] Ramin SM, Gambling DR, Lucas MJ, Sharma SK, Sidawi JE, Leveno KJ. Randomized trial of epidural versus intravenous analgesia during labor. Obstet Gynecol. 1995 Nov;86(5):783-9. doi: 10.1016/0029-7844(95)00269-w. PMID 7566849
- [Background] Sharpe EE, Arendt KW. Epidural Labor Analgesia and Maternal Fever. Clin Obstet Gynecol. 2017 Jun;60(2):365-374. doi: 10.1097/GRF.0000000000000270. PMID 28079555
- [Background] Kovo M, Schreiber L, Ben-Haroush A, Shor S, Golan A, Bar J. Intrapartum fever at term: clinical characteristics and placental pathology. J Matern Fetal Neonatal Med. 2012 Aug;25(8):1273-7. doi: 10.3109/14767058.2011.629248. Epub 2011 Nov 4. PMID 21992451
- [Background] Perlman JM. Maternal fever and neonatal depression: preliminary observations. Clin Pediatr (Phila). 1999 May;38(5):287-91. doi: 10.1177/000992289903800506. PMID 10349526
- [Background] Burgess APH, Katz JE, Moretti M, Lakhi N. Risk Factors for Intrapartum Fever in Term Gestations and Associated Maternal and Neonatal Sequelae. Gynecol Obstet Invest. 2017;82(5):508-516. doi: 10.1159/000453611. Epub 2017 Jan 20. PMID 28103590
- [Background] Dior UP, Kogan L, Calderon-Margalit R, Burger A, Amsallem H, Elchalal U, Eventov-Friedman S, Ergaz Z, Ezra Y. The association of maternal intrapartum subfebrile temperature and adverse obstetric and neonatal outcomes. Paediatr Perinat Epidemiol. 2014 Jan;28(1):39-47. doi: 10.1111/ppe.12090. Epub 2013 Oct 10. PMID 24118104
- [Background] Dior UP, Kogan L, Eventov-Friedman S, Gil M, Bahar R, Ergaz Z, Porat S, Calderon-Margalit R. Very High Intrapartum Fever in Term Pregnancies and Adverse Obstetric and Neonatal Outcomes. Neonatology. 2016;109(1):62-8. doi: 10.1159/000440938. Epub 2015 Nov 5. PMID 26536344
- [Background] Lieberman E, Eichenwald E, Mathur G, Richardson D, Heffner L, Cohen A. Intrapartum fever and unexplained seizures in term infants. Pediatrics. 2000 Nov;106(5):983-8. doi: 10.1542/peds.106.5.983. PMID 11061764
- [Background] Abdullahi H, Satti M, Rayis DA, Imam AM, Adam I. Intra-partum fever and cerebral palsy in Khartoum, Sudan. BMC Res Notes. 2013 Apr 24;6:163. doi: 10.1186/1756-0500-6-163. PMID 23618409
- [Background] Goodlin RC, Chapin JW. Determinants of maternal temperature during labor. Am J Obstet Gynecol. 1982 May 1;143(1):97-103. doi: 10.1016/0002-9378(82)90689-5. PMID 7081319
- [Background] Glosten B, Savage M, Rooke GA, Brengelmann GL. Epidural anesthesia and the thermoregulatory responses to hyperthermia--preliminary observations in volunteer subjects. Acta Anaesthesiol Scand. 1998 Apr;42(4):442-6. doi: 10.1111/j.1399-6576.1998.tb05139.x. PMID 9563864
- [Background] Goetzl L. Epidural analgesia and maternal fever: a clinical and research update. Curr Opin Anaesthesiol. 2012 Jun;25(3):292-9. doi: 10.1097/ACO.0b013e3283530d7c. PMID 22473213
- [Background] Segal S. Labor epidural analgesia and maternal fever. Anesth Analg. 2010 Dec;111(6):1467-75. doi: 10.1213/ANE.0b013e3181f713d4. Epub 2010 Sep 22. PMID 20861420
- [Background] Chen X, Ni X, Zhang Y, Liu H, Liu Z. The association of labor epidural analgesia with low concentration of ropivacaine and maternal fever: A retrospective study. J Clin Anesth. 2020 Oct;65:109613. doi: 10.1016/j.jclinane.2019.09.007. Epub 2020 May 15. No abstract available. PMID 32422544
- [Background] Zhou X, Li J, Deng S, Xu Z, Liu Z. Ropivacaine at different concentrations on intrapartum fever, IL-6 and TNF-alpha in parturient with epidural labor analgesia. Exp Ther Med. 2019 Mar;17(3):1631-1636. doi: 10.3892/etm.2018.7121. Epub 2018 Dec 20. PMID 30783430
- [Background] Wang T, Lu Y, Zhou P, Huang S, Yu X. A Randomized Controlled Comparison of Epidural Analgesia Onset Time and Adverse Reactions During Labor With Different Dose Combinations of Bupivacaine and Sufentanil. Clin J Pain. 2020 Aug;36(8):612-617. doi: 10.1097/AJP.0000000000000837. PMID 32349005
- [Background] Boudou M, Teissedre F, Walburg V, Chabrol H. [Association between the intensity of childbirth pain and the intensity of postpartum blues]. Encephale. 2007 Oct;33(5):805-10. doi: 10.1016/j.encep.2006.10.002. French. PMID 18357852
- [Background] Ding T, Wang DX, Qu Y, Chen Q, Zhu SN. Epidural labor analgesia is associated with a decreased risk of postpartum depression: a prospective cohort study. Anesth Analg. 2014 Aug;119(2):383-392. doi: 10.1213/ANE.0000000000000107. PMID 24797120
- [Background] Suhitharan T, Pham TP, Chen H, Assam PN, Sultana R, Han NL, Tan EC, Sng BL. Investigating analgesic and psychological factors associated with risk of postpartum depression development: a case-control study. Neuropsychiatr Dis Treat. 2016 Jun 9;12:1333-9. doi: 10.2147/NDT.S105918. eCollection 2016. PMID 27354803
- [Background] Liu ZH, He ST, Deng CM, Ding T, Xu MJ, Wang L, Li XY, Wang DX. Neuraxial labour analgesia is associated with a reduced risk of maternal depression at 2 years after childbirth: A multicentre, prospective, longitudinal study. Eur J Anaesthesiol. 2019 Oct;36(10):745-754. doi: 10.1097/EJA.0000000000001058. PMID 31356375